CLINICAL TRIAL: NCT07176624
Title: The Effect of Reducing Enteral Nutrition Before Prone Positioning on Clinical Outcomes in Mechanically Ventilated ARDS Patients: A Multicenter Randomized Controlled Trial (The PRE-VAIL Study)
Brief Title: The PRE-VAIL Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The PRE-VAIL Study
Record Dates: First submitted 2025-07-30; First posted 2025-09-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-08

CONDITIONS: ARDS (Moderate or Severe); Prone Position; Enteral Nutrition Feeding; Intensive Care Unit (ICU) Admission
Keywords: ARDS; Mechanical ventilation; Prone position; Enteral nutrition; Gastric retention; Clinical outcome
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral nutrition reduction group (Experimental): Before the prone position, the gastric contents are aspirated with a syringe, and the dose of enteral nutrition reduction is determined based on the different amounts of gastric residue. If the residual volume in the stomach is less than 200ml, the enteral nutrition intake will be reduced by one third. Gastric residual volume 200-500ml: Reduce enteral nutrition by half. If the residual gastric volume is greater than 500ml: Stop enteral nutrition and consider post-pyloric feeding
  Interventions: Procedure: Enteral nutrition is reduced before the prone position
- Conventional feeding group (No Intervention): Do not reduce the feeding speed before the prone position and continue to feed at the original speed

INTERVENTIONS:
Procedure: Enteral nutrition is reduced before the prone position — Before the prone position, the gastric contents are aspirated with a syringe, and the dose of enteral nutrition reduction is determined based on the different amounts of gastric residue. If the residual volume in the stomach is less than 200ml, the enteral nutrition intake will be reduced by one third. Gastric residual volume 200-500ml: Reduce enteral nutrition by half. If the residual gastric volume is greater than 500ml: Stop enteral nutrition and consider post-pyloric feeding
  Arms: Enteral nutrition reduction group

SUMMARY:
During the prone position, there may be an increase in intragastric pressure. The investigators focus on a scientific question: Whether reducing enteral nutrition before the prone position will benefit patients with severe mechanically ventilated acute respiratory distress syndrome (ARDS).

The experimental group had the enteral nutrition dose reduced before the prone position, while the control group did not have the enteral nutrition dose reduced

DETAILED DESCRIPTION:
During the prone position, there may be an increase in intragastric pressure. The investigators focus on a scientific question: Whether reducing enteral nutrition before the prone position will benefit patients with severe mechanically ventilated ARDS.

The experimental group had the enteral nutrition dose reduced before the prone position, while the control group did not have the enteral nutrition dose reduced

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Within 24 hours of admission to the ICU, one or more organ systems have failed (the Sequential Organ Failure Assessment (SOFA) score of any single organ system is ≥2)
* Meet the diagnostic criteria for moderate/severe ARDS (even after optimizing the ventilation Settings, the oxygenation index is still < 150mmHg and PEEP is still ≥5 cm H2O)
* It is expected to stay in the ICU for more than 48 hours

Exclusion Criteria:

* There are contraindications for the prone position
* There are contraindications for EN, preventing the initiation of early EN (≤48 hours)
* Expected to die within 48 hours
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Estimated)
Dates: Start 2025-09-14 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2028-02-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of gastric retention during prone position | Acute stage of critical illness (within 7 days of Intensive Care Unit (ICU))
  The incidence of gastric retention (with a single gastric residual volume > 200ml) during prone position.

SECONDARY OUTCOMES:
The frequency of gastric retention during the prone position | Acute stage of critical illness (within 7 days of ICU)
  The number of times of gastric retention (with a single gastric residual volume > 200ml) per unit time during prone position (times per day)
The incidence of diarrhea during ICU stay | Acute stage of critical illness (within 7 days of ICU)
  Having three or more loose or liquid stools per day, with a stool weight greater than 200-250g/d (or more than 250ml/d)
EN interruption rate | Acute stage of critical illness (within 7 days of ICU)
  High gastric residual volume (single dose > 500ml) or serious gastrointestinal adverse events lead to the need to suspend EN administration
The incidence of Ventilator-associated pneumonia (VAP) among the participants | During the length of stay in the ICU (from day 1 to a maximum of 28 days)
  Pulmonary infectious inflammation that occurs 48 hours after the end of ventilator treatment is a type of hospital-acquired pneumonia
Nutrition compliance rate | The seventh day in the ICU
  Whether the patient reached 80% of the nutritional (calories: 25kcal/kg/day and protein :1.3g/kcal) target on the 7th day of hospitalization in the ICU
Gastric antral cross-sectional area (ACSA) measured by ultrasound after the end of prone positioning | After each prone position during the ICU stay
  The ultrasound cross-sectional area of the antrum of the stomach after adjusting to the normal position at the end of the prone position
Length of stay in the ICU | During the length of stay in the ICU (from day 1 to a maximum of 180 days)
  The number of days spent in the ICU
ICU mortality | During the length of stay in the ICU (from day 1 to a maximum of 180 days)
  Whether there was death during the ICU stay
28-day mortality | Day 28 after being admitted to the ICU
  Whether the patient died on the 28th day after being admitted to the ICU
90-day mortality | The 90th day after being admitted to the ICU
  Whether the patient died on the 90th and 180th days after being admitted to the ICU
180-day mortality | Day 180 after being admitted to the ICU
  Whether the patient died on the 180th day after being admitted to the ICU
The incidence of gastric retention during ICU stay | Within 1 to 7 days of hospitalization in the ICU
  The incidence of gastric retention within 7 days of ICU hospitalization (The single gastric residual volume is greater than 200ml)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available upon reasonable request. Researchers interested in obtaining the data should contact the corresponding author with a clear statement of the purpose of data access. The corresponding author will evaluate the request and determine whether access can be granted to part of the de-identified dataset.